CLINICAL TRIAL: NCT04308265
Title: Does the Scoring System Affect the Surgery Timing in Acute Calculous Cholecystitis?
Brief Title: Scoring System in Acute Calculous Cholecystitis
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, principal investigators, Konya Meram State Hospital
Other Study IDs: Department of general surgery
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Acute cholecystitis is a common disease in the daily practice of general surgery. There are various methods in the treatment of this disease, such as early cholecystectomy, medical treatment, six weeks later cholecystectomy and cholecystostomy. However, it is not satisfied with objective criteria that these methods are selected according to which patient groups. With this observational-prospective study, the benefit of first visit scoring on 'which of the treatment options will be most suitable for the patient' will be investigated. Thus, rare but severe complications of cholecystectomy can be prevented.

DETAILED DESCRIPTION:
Acute cholecystitis refers to acute inflammation of the gallbladder, and why it is often gallstones. Gallstones are seen in western society with about 10% frequency, while 80% of them are asymptomatic. Acute cholecystitis accounts for 1-3% of those with symptomatic gallstones.

Acute cholecystitis is a table characterized by right upper quadrant pain (in the inflammatory pain pattern and continuous), defensiveness in the right upper quadrant (murphy manifestation is positive or not), and an increase in inflammatory response parameters (such as fever, white blood cell, and CRP elevation). Biliary scintigraphy, called the HIDA scan, is the gold standard method in diagnosis. However, due to the difficulty and cost of application, ultrasonography is used in the routine application in diagnosis. It is valuable that gallstones and gallbladder walls are thicker than 4 mm in ultrasonography. However, pericholecystic fluid is a more valuable finding and is rare.

In the treatment of acute cholecystitis, the patient's hospitalization, limiting oral food intake, IV hydration, NSAID, and antibiotic treatment is the main conservative approaches. While these patients were admitted to the hospital in the first 72 hours from the onset of symptoms, early cholecystectomy is recommended. If they arrive later, interval cholecystectomy is recommended after 6-8 weeks. Laparoscopic cholecystectomy is recommended for all operations. However, the choice of surgical treatment is determined by the surgeon, according to the patient. More precise and objective criteria are needed to contribute to this choice.

In a study comparing early cholecystectomy and delayed cholecystectomy, intraoperative and postoperative complications were more common in early cholecystectomy than interval cholecystectomy. Still, early cholecystectomy had better results in terms of cost and hospital stay. There are many studies in the literature comparing early and late cholecystectomy. In these studies, the selection criteria of patients are different in all of them.

Finally, it was emphasized that a retrospective scoring study conducted in Germany could be successful in patient selection.

In conclusion, the debate on treatment choices of patients with acute cholecystitis continues. Recent publications in the literature on the development of scoring systems for these patients draw attention, so investigators want to investigate the effectiveness of a scoring system in which patients are evaluated in many ways.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and Radiologically diagnosed with acute cholecystitis
* be over 18 years old

Exclusion Criteria:

* Being under the age of 18
* getting pregnant
* Acute pancreatitis, cholangitis or choledochal stone with acute cholecystitis
* Having a previous history of upper abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital for acute cholecystitis older than 18 years will constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-03-07 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
cut off value | Three months
  After entering the patients' data entries and scoring points, ROC analysis will be done with the SPSS program. The resulting cut off value is given to us; It will provide information about which patients to recommend early cholecystectomy, which patients should seek medical treatment and other solutions.
  Values above the cut-off value to be analyzed will be considered bad value. If values above the cut off value are found, surgery will not be preferred.
The score will be determined. | Three months
  A score will be determined with the scoring system created using the history, history information, hemogram, biochemistry tests, ultrasonography findings of the patients admitted to the study, and the height and bodyweight of the patients.
  Scoring will be created using the following information;
  * Diabetes Mellitus story
  * White Blood Cell
  * C Reactive Protein (CRP)
  * Wall thickness of gall bladder
  * Pericholecystic Fluid
  * Acute Cholecystitis Attack Number
  * Pain start time (hours)
  * AGE
  * GENDER
  * Body Mass Index

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozkardes AB, Tokac M, Dumlu EG, Bozkurt B, Ciftci AB, Yetisir F, Kilic M. Early versus delayed laparoscopic cholecystectomy for acute cholecystitis: a prospective, randomized study. Int Surg. 2014 Jan-Feb;99(1):56-61. doi: 10.9738/INTSURG-D-13-00068.1. PMID 24444271
- [Result] Ambe PC, Papadakis M, Zirngibl H. A proposal for a preoperative clinical scoring system for acute cholecystitis. J Surg Res. 2016 Feb;200(2):473-9. doi: 10.1016/j.jss.2015.09.010. Epub 2015 Sep 9. PMID 26443188